CLINICAL TRIAL: NCT00778986
Title: Effects of Remote Patient Monitoring on Heart Failure Management: A Randomized Controlled Trial
Brief Title: Effects of Remote Patient Monitoring on Heart Failure Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Heather Ross, University Health Network
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HF-RPM-UHN
Record Dates: First submitted 2008-10-23; First posted 2008-10-24 (Estimated); Last update posted 2010-09-30 (Estimated); Status verified 2010-09

CONDITIONS: Heart Failure
Keywords: heart failure; remote patient monitoring; telemonitoring; home monitoring; randomized controlled trial; self care
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- remote monitoring (Experimental): group of patients that will be using the heart failure remote patient monitoring system in addition to the usual care they receive at the University Health Network Heart Failure Clinic
  Interventions: Device: heart failure remote patient monitoring system
- control (No Intervention): group of patients provided with usual care at the University Health Network Heart Failure Clinic

INTERVENTIONS:
Device: heart failure remote patient monitoring system — remote monitoring of weight, blood pressure, ECG, and symptoms
  Arms: remote monitoring

SUMMARY:
The purpose of this randomized controlled trial is to determine the effects of a user-centric remote patient monitoring system on heart failure management. Patients attending a Heart Failure Clinic will monitor their weight, blood pressure, ECG, and symptoms at home. The hypothesis is that the remote monitoring system will improve heart failure outcomes through increased self-care and improved clinical management.

DETAILED DESCRIPTION:
Poor management of heart failure (HF) has added to the high costs and negative health outcomes from this chronic illness, including frequent hospitalization. HF patients require close monitoring to detect worsening health and to optimize their treatment. However, many patients visit their HF clinicians only once every few months, and perform minimal or no self-monitoring.

Remote patient monitoring is a potential tool to help clinicians and the patients better manage HF. A remote patient monitoring system (home monitoring of vital signs and symptoms) that has been developed with extensive clinician and patient input and testing, will be studied to determine its effects on HF management. Half of one hundred patients from the University Health Network Heart Failure Clinic will be randomly placed into the remote monitoring (RM) group and the other half will be in the control group. Patients in the RM group will monitor their weight, blood pressure, ECG, and symptoms at home for 6 months. This information will be automatically sent from the medical devices wirelessly through Bluetooth to a mobile phone, which will send the information to the data servers. Both clinicians and patients will have access to the data. Patients will get automated reminder telephone calls if they do not take the number of measurements prescribed by their doctors.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Heart Failure (NYHA Class II-IV)
* Out-patients attending the University Health Network Heart Failure Clinic
* English-speaking and able to read English
* 18 years old or over

Exclusion Criteria:

* Awaiting heart transplantation
* Not expected to survive over a year (as determined by their cardiologist)
* Unable to read text on a mobile phone due to vision disability
* Unable to self-care due to anxiety, depression, or decreased cognitive function
* Lack of manual dexterity to accurately press buttons on the mobile phone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-03; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Brain Natriuretic Peptide values | Baseline, 6 months
Self-care practices measured through Self-Care of Heart Failure Index scores and interviews | baseline, 6 months
Health related quality of life measured through the Minnesota Living with Heart Failure Questionnaire scores and interviews | baseline, 6 months

SECONDARY OUTCOMES:
Number of hospitalizations and days in hospital | 6 months comparison between intervention and control groups
Number of Emergency Department visits | 6 month comparison between intervention and control groups
All cause mortality | 6 month comparison between intervention and control groups
Number of Heart Failure Clinic visits | 6 month comparison between intervention and control groups

CONTACTS AND LOCATIONS:
Overall Officials: Heather J Ross, MD, MHSc, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Seto E, Leonard KJ, Cafazzo JA, Barnsley J, Masino C, Ross HJ. Developing healthcare rule-based expert systems: case study of a heart failure telemonitoring system. Int J Med Inform. 2012 Aug;81(8):556-65. doi: 10.1016/j.ijmedinf.2012.03.001. Epub 2012 Mar 31. PMID 22465288
- [Derived] Seto E, Leonard KJ, Cafazzo JA, Barnsley J, Masino C, Ross HJ. Mobile phone-based telemonitoring for heart failure management: a randomized controlled trial. J Med Internet Res. 2012 Feb 16;14(1):e31. doi: 10.2196/jmir.1909. PMID 22356799